CLINICAL TRIAL: NCT00446511
Title: An Extension to Study Protocol CVAL489K2302 to Evaluate the Long Term Safety, Tolerability and Efficacy of Valsartan in Children 6 to 17 Years of Age With Hypertension, Versus Enalapril Treatment for 14 Weeks, or Combined With Enalapril Versus Enalapril for 66 Weeks in Chronic Kidney Disease Patients.
Brief Title: Extension Study to Assess Long Term Safety, Tolerability, and Efficacy of Valsartan and Enalapril Combined and Alone in Children With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAL489K2302E1
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: children; pediatrics; high blood pressure; hypertension; valsartan; enalapril
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CKD patients: Valsartan+enalapril (Experimental)
  Interventions: Drug: Valsartan; Drug: Enalapril
- CKD patients: Enalapril (Active Comparator)
  Interventions: Drug: Enalapril; Drug: placebo matched to valsartan
- Non-CKD patients: Valsartan (Experimental)
  Interventions: Drug: Valsartan; Drug: placebo matched to enalapril
- Non-CKD patients: Enalapril (Active Comparator)
  Interventions: Drug: Enalapril; Drug: placebo matched to valsartan

INTERVENTIONS:
Drug: Valsartan — Valsartan (80, 160, and 320 mg, weight stratified). All study medications were taken orally once daily, at approximately the same time each day, with or without food.
  Arms: CKD patients: Valsartan+enalapril; Non-CKD patients: Valsartan
Drug: Enalapril — Enalapril (10, 20, and 40 mg, weight stratified). All study medications were taken orally once daily, at approximately the same time each day, with or without food.
  Arms: CKD patients: Enalapril; CKD patients: Valsartan+enalapril; Non-CKD patients: Enalapril
Drug: placebo matched to enalapril — Placebo matched to enalapril. All study medications were taken orally once daily, at approximately the same time each day, with or without food.
  Arms: Non-CKD patients: Valsartan
Drug: placebo matched to valsartan — placebo matched to valsartan. All study medications were taken orally once daily, at approximately the same time each day, with or without food.
  Arms: CKD patients: Enalapril; Non-CKD patients: Enalapril

SUMMARY:
The purpose of this extension study is to compare the long-term safety of valsartan versus enalapril, and the effectiveness of the combination of valsartan and enalapril versus enalapril alone in children with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of 12 weeks of double-blind treatment in core protocol CVAL489K2302.
* Patients participating in study CVAL489K2302 who may have discontinued prematurely due to uncontrolled hypertension defined as MSSBP > 20%, but < 25% above the 95th percentile for age, gender, and height after visit 5, qualifies a patient for entry into this extension study.

Exclusion Criteria:

* Renal artery stenosis.
* Current diagnosis of heart failure (NYHA Class II-IV).
* Second or third degree heart block without a pacemaker.
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia.
* Clinically significant valvular heart disease.
* Patient that demonstrates clinically significant ECG abnormalities other than those associated with left ventricular hypertrophy and AV block controlled with a pacemaker.
* Previous solid organ transplantation except renal, liver or heart transplantation. Renal, liver or heart transplant must have occurred at least 6 months prior to enrollment. Patient must be on stable doses of immunosuppressive therapy for 3 months and deemed clinically stable by the investigator.
* Patients who experienced any adverse events considered serious and drug related in protocol CVAL489K2302.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (9):
- Sites in USA, East Hanover, New Jersey, United States
- Sites in Belgium, Belgium, Belgium
- Sites in France, France, France
- Sites in Germany, Germany, Germany
- Sites in Hungary, Hungary, Hungary
- Sites in India, India, India
- Sites in Italy, Italy, Italy
- Sites in Poland, Poland, Poland
- Sites in Turkey, Turkey, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- CKD Patients: Valsartan+Enalapril: Chronic kidney disease (CKD) patients assigned to valsartan in the core study received combination therapy of valsartan and enalapril in the extension: Valsartan+enalapril (80/10, 160/20, 320/40 mg, weight stratified). All study medications were taken orally once daily, at approximately the same time each day, with or without food.
- CKD Patients: Enalapril: Chronic kidney disease (CKD) patients assigned to enalapril in the core study received enalapril and valsartan placebo in the extension: Enalapril (10, 20, 40, weight stratified) and matching placebo to valsartan (80, 160, 320 mg). All study medications were taken orally once daily, at approximately the same time each day, with or without food.
- Non-CKD Patients: Valsartan: Non-chronic kidney disease (CKD) patients assigned to valsartan in the core study continued their valsartan monotherapy treatment in the extension: Valsartan (80, 160, 320 mg, weight stratified)+enalapril placebo. All study medications were taken orally once daily, at approximately the same time each day, with or without food.
- Non-CKD Patients: Enalapril: Non-chronic kidney disease (CKD) patients assigned to enalapril in the core study continued their enalapril monotherapy treatment in the extension: Enalapril (10, 20, 40, weight stratified)+valsartan placebo. All study medications were taken orally once daily, at approximately the same time each day, with or without food.
Period: Overall Study
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Started | 21 | 17 | 103 | 109
Completed | 11 | 15 | 96 | 103
Not Completed | 10 | 2 | 7 | 6
Not completed — Adverse Event | 7 | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Administrative Problems | 3 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril | Total
Number analyzed (Participants) | 21 | 17 | 103 | 109 | 250
Age Continuous [Mean (Standard Deviation); unit: years] | 11.4 (3.40) | 12.1 (3.07) | 13.1 (2.75) | 13.3 (2.81) | 13.0 (2.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 41 | 27 | 81
  Male | 13 | 12 | 62 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Time Frame: Start of extension (week 13) to end of study (Week 26 in non-CKD patients and Week 50 in CKD patients)
Population: Extension safety population
Measure: Number; unit: Participants
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Number analyzed (Participants) | 21 | 17 | 103 | 109
Participants | 16 | 11 | 51 | 53

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to Week 26
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using a calibrated standard sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit. A negative number indicates lowered blood pressure.
Time Frame: Core Baseline (Week 0) to Week 26
Population: Extension ITT population: All patients that had both baseline and at least 1 post-Week 12 assessment of any efficacy variable (sitting systolic/diastolic BP) during the extension. Baseline is the Week 0 value. Extension endpoint is the Week 26 or last observation after the core endpoint but before Week 26 carried forward value.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Number analyzed (Participants) | 21 | 17 | 103 | 108
mmHg | -20.4 (11.48) | -11.7 (9.55) | -7.5 (8.47) | -7.2 (8.99)

3. Secondary Outcome: Percentage of Non-CKD Patients Achieving Systolic and Diastolic BP Control at Week 26
Description: Systolic and diastolic blood pressure (BP) control was defined as msSBP and msDBP < 95th percentile for gender, age, and height. After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using a calibrated standard sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit.
Time Frame: Week 26
Population: The extension ITT population consisted of all extension patients that had both baseline and at least one post-Week 12 assessment of any efficacy variable (sitting systolic/diastolic blood pressure) during the extension. Patients were analyzed according to the treatment they were assigned to at the beginning of their extension.
Measure: Number; unit: Percentage of patients
Groups:
- Non-CKD Patients: Valsartan: All non-CKD patients assigned to valsartan in the core study (CVAL489K2302) continued their monotherapy treatment of valsartan 80/160/320 mg stratified by weight.
- Non-CKD Patients: Enalapril: All non-CKD patients assigned to enalapril in the core study (CVAL489K2302) continued their monotherapy treatment of enalapril 10/20/40 mg stratified by weight.
Arm/Group | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Number analyzed (Participants) | 103 | 108
Percentage of patients
  Systolic BP control | 66.0 | 63.0
  Diastolic BP control | 95.1 | 91.7

4. Secondary Outcome: Change From Baseline in Post-dosing 24-hour Mean Systolic and Diastolic Ambulatory Blood Pressure at Week 20
Description: 24-hour ambulatory blood pressure monitoring (ABPM) was conducted once during the extension in a subset of patients at selected centers. For all patients who completed a qualifying ABPM at baseline, an ABPM was to be performed at Week 20. The ABPM monitor was placed on the non-dominant arm.
Time Frame: Core Baseline (Week 0) to Week 20
Population: ABPM population: All ITT patients who received the 24-hour ambulatory blood pressure monitoring (ABPM) measurements at both baseline and Week 20. Patients were excluded if their baseline ABPM was measured after active treatment dose (considered invalid baseline).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Number analyzed (Participants) | 5 | 2 | 10 | 21
mmHg
  Systolic BP | -23.3 (11.60) | -0.3 (14.42) | -11.5 (7.81) | -4.1 (11.49)
  Diastolic BP | -17.8 (3.20) | 2.9 (10.81) | -12.2 (6.60) | -4.5 (7.59)

5. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to Week 26
Description: as for outcome 2
Time Frame: Core Baseline (Week 0) to Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CKD Patients: Valsartan+Enalapril | CKD Patients: Enalapril | Non-CKD Patients: Valsartan | Non-CKD Patients: Enalapril
Number analyzed (Participants) | 21 | 17 | 103 | 108
mmHg | -23.6 (10.79) | -18.2 (9.51) | -11.6 (9.74) | -10.2 (9.70)

ADVERSE EVENTS:
Time Frame: Start of extension (week 13) to end of study (Week 26 in non-CKD patients and Week 50 in CKD patients).
Arm/Group | CKD Patients: Valsartan+Enalapril | Non-CKD Patients: Valsartan | CKD Patients: Enalapril | Non-CKD Patients: Enalapril
Serious Adverse Events (participants affected / at risk) | 7/21 | 1/103 | 0/17 | 2/109
Other Adverse Events (participants affected / at risk) | 14/21 | 25/103 | 11/17 | 42/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CKD Patients: Valsartan+Enalapril (N=21) | Non-CKD Patients: Valsartan (N=103) | CKD Patients: Enalapril (N=17) | Non-CKD Patients: Enalapril (N=109)
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Synostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CKD Patients: Valsartan+Enalapril (N=21) | Non-CKD Patients: Valsartan (N=103) | CKD Patients: Enalapril (N=17) | Non-CKD Patients: Enalapril (N=109)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Pyrexia (General disorders) | 3 | 5 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 6 | 1 | 9
Pharyngitis (Infections and infestations) | 2 | 7 | 2 | 11
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 11 | 1 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was prolonged from 14 to 66 wks for CKD patients only. Most CKD patients completed the initial 14 wk extension period prior to amendment approval and the study was terminated prematurely with 3 CKD patients progressing to a maximum of Visit 13.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.